CLINICAL TRIAL: NCT00545883
Title: An Epidemiological, Observational Study to Describe Symptom Control and Impact on Daily Life of GERD in Patients With Erosive Gastroesophageal Reflux Disease.
Brief Title: Impact of GERD on Daily Life (NIS)
Acronym: Alegria
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-GBE-NEX-2006/1
Record Dates: First submitted 2007-10-15; First posted 2007-10-17 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: GERD
Keywords: GERD; esophagitis; PPI
MeSH Terms: conditions — Gastroesophageal Reflux; Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to gather epidemiological data in a population of GERD patients in primary care with a history of erosive esophagitis (less than or equal to 3 years).

ELIGIBILITY:
Inclusion Criteria:

* Patients with erosive esophagitis (endoscopical findings according to the Los Angeles Classification; grade A-D) currently not treated with a proton pump inhibitor, for whom the general practitioner (GP) has decided to initiate or change the treatment for GERD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary & Specialty care units
Sampling Method: Non-Probability Sample
Enrollment: 2001 (Actual)
Dates: Start 2006-06; Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
To gather epidemiological data in a population of GERD patients | After collection of all questionnaires

SECONDARY OUTCOMES:
To evaluate the added value of a new patient questionnaire (GERD Impact Scale) as a useful tool for the initial and long-term management of GERD patients: determination of the appropriate treatment and evaluation of the response to treatment. | After collection of all questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: E. Louis, PR, Principal Investigator — ULG
Locations (112):
- Belgium (112):
  - Research Site, Aarschot
  - Research Site, Aartselaar
  - Research Site, Alken
  - Research Site, Angleur
  - Research Site, Antwerp
  - Research Site, Balen
  - Research Site, Berchem
  - Research Site, Beringen
  - Research Site, Beyne-Heusay
  - Research Site, Boechout
  - Research Site, Boirs
  - Research Site, Boom
  - Research Site, Borgerhout
  - Research Site, Bornem
  - Research Site, Brussels
  - Research Site, Chênée
  - Research Site, Court-Saint-Étienne
  - Research Site, Deurne
  - Research Site, Diegem
  - Research Site, Diest
  - Research Site, Dilbeek
  - Research Site, Duffel
  - Research Site, Eindhout
  - Research Site, Ekeren
  - Research Site, Essen
  - Research Site, Flémalle
  - Research Site, Fléron
  - Research Site, Geel
  - Research Site, Genk
  - Research Site, Gooik
  - Research Site, Grand-Rechain
  - Research Site, Grâce-Hollogne
  - Research Site, Grivegnée
  - Research Site, Grobbendonk
  - Research Site, Groot-Biigaarden
  - Research Site, Halen
  - Research Site, Hannut
  - Research Site, Herentals
  - Research Site, Herenthout
  - Research Site, Hermalle-sous-Huy
  - Research Site, Herselt
  - Research Site, Herstal
  - Research Site, Herve
  - Research Site, Heusden-Zolder
  - Research Site, Hoboken
  - Research Site, Hoeilaart
  - Research Site, Houthalen-Helchteren
  - Research Site, Huy
  - Research Site, Itegem
  - Research Site, Ivoz-Ramet
  - Research Site, Jodoigne
  - Research Site, Keerbergen
  - Research Site, Kortrijk-Dutsel
  - Research Site, Landen
  - Research Site, Lasne
  - Research Site, Leefdaal
  - Research Site, Leopoldsburg
  - Research Site, Liederkerke
  - Research Site, Lier
  - Research Site, Liège
  - Research Site, Lommel
  - Research Site, Londerzeel
  - Research Site, Louveigné
  - Research Site, Maasmechelen
  - Research Site, Mechelen
  - Research Site, Merksem
  - Research Site, Munsterbilzen
  - Research Site, Niel
  - Research Site, Noordewijk
  - Research Site, Olen
  - Research Site, Oostmalle
  - Research Site, Overpelt
  - Research Site, Paal-Beringen
  - Research Site, Pellaines
  - Research Site, Peutie
  - Research Site, Pulle
  - Research Site, Putte
  - Research Site, Puurs
  - Research Site, Reet
  - Research Site, Retie
  - Research Site, Retinne
  - Research Site, Riemst
  - Research Site, Rijkhoven
  - Research Site, Rixensart
  - Research Site, Roosdaal
  - Research Site, Schelle
  - Research Site, Schilde
  - Research Site, Schulen-herk-de-stad
  - Research Site, Seraing
  - Research Site, Spouwen
  - Research Site, Stabroek
  - Research Site, Steenokkerzeel
  - Research Site, Ternat
  - Research Site, Tessenderlo
  - Research Site, Tienen
  - Research Site, Tollembeek
  - Research Site, Tongeren
  - Research Site, Vierset-Barse
  - Research Site, Viller-le-Temple
  - Research Site, Vilvoorde
  - Research Site, Walem
  - Research Site, Wambeek
  - Research Site, Weerde
  - Research Site, Wespelaar
  - Research Site, Westerlo
  - Research Site, Westmeerbeek
  - Research Site, Willebroek
  - Research Site, Wilrijk
  - Research Site, Wolvertem
  - Research Site, Zandhoven
  - Research Site, Zemst
  - Research Site, Zichem